CLINICAL TRIAL: NCT01078350
Title: Consent for Obtaining Additional Tissue at the Time of a Diagnostic Biopsy
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: BANKPEDSTS0001; 80003; SU-11052007-794 (Other: Stanford)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma; Hodgkin Disease
Keywords: Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissues sample

INTERVENTIONS:
Procedure: tumor tissue aspiration
Procedure: phlebotomy

SUMMARY:
This study is designed to collect tissue samples that may aid in the treatment and learning about various oncology diagnosis.

DETAILED DESCRIPTION:
The purpose of this study is to provide a mechanism to obtain tissue specimens to be used for experimental studies before the exact histologic diagnosis is known.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are having a tissue procedure done as part of their standard oncology work-up will be eligible to be consented on this study.

Exclusion Criteria:

* None.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects who are having a tissue procedure done as part of their standard oncology work-up will be eligible to be consented on this study.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2015-12-04 (Actual)

PRIMARY OUTCOMES:
Further analysis | at collection time

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Neyssa Marina, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States